CLINICAL TRIAL: NCT05051033
Title: Percutaneous or Surgical Repair In Mitral Prolapse And Regurgitation for ≥60 Year-olds (PRIMARY)
Acronym: PRIMARY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Annetine Gelijns (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Annetine Gelijns, Chair, Department of Population Health Science & Policy Edmond A. Guggenheim Professor of Health Policy Co-Director, InCHOIR, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-01246; 5U01HL088942 (NIH)
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Mitral Valve Regurgitation
Keywords: surgical mitral valve repair; transcatheter edge-to-edge repair
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Intervention Model Description: Eligible and consented patients will be randomized 1:1 to a TEER versus surgical repair. Patient randomization will be stratified by clinical site and by surgical risk profile, namely low, intermediate, and high surgical risk. Primary effectiveness will be analyzed by intention-to-treat; that is, the patients will be grouped by their assignment at randomization whether or not they actually received the treatment to which they were assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Surgical mitral valve repair (Active Comparator): Patients who are randomized to the surgical arm will undergo mitral surgery.
  Interventions: Procedure: Mitral valve repair
- Transcatheter edge-to-edge repair (Active Comparator): In the transcatheter edge-to-edge repair arm, patients will be treated with a commercially-approved edge-to-edge mitral repair device.
  Interventions: Device: Transcatheter edge-to-edge repair

INTERVENTIONS:
Procedure: Mitral valve repair — Patients who are randomized to the surgical arm will undergo mitral surgery. Mitral surgery will be conducted using general anesthesia and cardiopulmonary bypass. Mitral surgery may be performed via a sternotomy or a right thoracotomy approach with or without robotic assistance. Standard techniques commonly include a ring or band annuloplasty to correct and prevent annular dilatation; leaflet prolapse and redundancy may be corrected by leaflet resection techniques and / or chordal reconstruction.
  Other Names: Mitral valve surgery
  Arms: Surgical mitral valve repair
Device: Transcatheter edge-to-edge repair — Patients will be treated with a commercially-approved edge-to-edge mitral repair device. The steerable guide catheter (guide) is inserted into the femoral vein and advanced across the inter-atrial septum using image guided puncture. Fluoroscopic and echocardiographic guidance will be used to visualize the devices and assess the repair. The guide is positioned over the MV and the clip/clasp delivery system is inserted into the guide and positioned over the MV in accordance with the manufacturer's instructions. The delivery catheter is advanced until the clip/clasp emerges from the tip of the guide into the left atrium. The catheter is manipulated using the control handle until the clip/clasp is correctly oriented with respect to the line of coaptation of the mitral valve. The clip/clasp is opened, and advanced across the mitral valve into the left ventricle then pulled back to grasp the leaflets.
  Other Names: TEER
  Arms: Transcatheter edge-to-edge repair

SUMMARY:
This is a prospective, multicenter, open-label, randomized trial comparing mitral valve (MV) transcatheter edge-to-edge repair (TEER) to surgical repair (1:1 ratio) in patients with primary, degenerative mitral regurgitation (MR). The trial will be conducted in the U.S., Canada, Germany, Spain, and the United Kingdom, and is designed as a strategy trial. Thus, all devices legally marketed for TEER of primary degenerative MR in a particular country are eligible to be used in this trial.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the long-term effectiveness and safety of MV TEER compared with surgical repair in patients with primary, degenerative MR. The secondary aim is to analyze the relationship between the adequacy of MR correction at one-year post intervention and longer-term clinical outcomes (death, heart failure hospitalizations/urgent care visits, valve re-interventions, and quality of life). The tertiary aim of this trial is to evaluate a range of patient-centered outcomes (quality of life, functional status, and discharge location) of transcatheter edge-to-edge MV repair compared with MV surgical repair in patients with primary, degenerative mitral regurgitation. This study is closely integrated with the PRIMARY Ancillary Substudy (NCT07103733)

The patient population for this trial consists of adult patients with severe, primary degenerative MR for whom the local heart team has verified that an indication for MV intervention is present and for whom both transcatheter edge-to-edge and surgical repair strategies are anatomically feasible.

Because the use of the commercial edge-to-edge mitral repair device in the U.S. is approved only in patients considered to be at prohibitive risk of MV surgery by a heart team, use of such devices in this trial is considered investigational by the FDA. As such, this trial will be conducted under an Investigational Device Exemption (IDE).

Outcomes will be measured from randomization over a period of 5 years post intervention. The estimated enrollment period is 36 months, and all patients will be followed from randomization for up to 10 years post intervention for particular endpoints. Long-term follow-up will include leveraging administrative datasets linked to clinical trial data.

ELIGIBILITY:
The patient population for this trial consists of adults with severe, primary degenerative MR for whom the local heart team has verified that an indication for MV intervention is present and for whom both transcatheter edge-to-edge and surgical repair strategies are anatomically feasible. Specific inclusion and exclusion criteria are listed below. All patients who meet eligibility criteria will be included in the study regardless of gender, race, or ethnicity.

Inclusion Criteria:

* Adult patients ≥60 years with moderately-severe or severe (3+ or 4+/4+) primary degenerative (Carpentier type II) MR defined by transthoracic echocardiography
* Clinical indication for MV intervention and anatomic candidate for both surgical MV repair and transcatheter edge-to-edge repair (TEER) per local heart team assessment with central eligibility committee verification
* Patients across the surgical risk spectrum (low, intermediate, and high risk) depending on local heart team assessment and central eligibility committee verification (see ACC/AHA 2020 guidelines for the management of patients with valvular heart disease)
* Patients with AF who meet an indication for a concomitant ablation procedure be included provided the local heart team and central eligibility committee decide they are eligible for both catheter-based and surgical ablation.
* Ability to perform 6-minute walk test (6MWT) and complete Kansas City Cardiomyopathy Questionnaire (KCCQ) instrument

Exclusion Criteria:

* Non-degenerative types of primary MR (e.g., cleft leaflet)
* Secondary or functional MR
* Hypertrophic obstructive cardiomyopathy
* Presence of an IVC filter or permanent pacing/ICD leads that would interfere with TEER per local heart team assessment
* Known allergic reactions to intravenous contrast
* Febrile illness within 30-days prior to randomization
* Any absolute contraindication to transesophageal echocardiography
* Any contraindication to systemic heparinization including active bleeding diatheses, and heparin induced thrombocytopenia
* Patients with CAD requiring revascularization
* Any prior mitral valve intervention or any prior repair of atrial septal defect
* Any prior MV intervention or any prior repair of atrial septal defect
* Need for any of the following concomitant procedures: aortic valve or aortic surgery, tricuspid valve surgery
* Need for any emergency intervention or surgery
* Active endocarditis
* Hemodynamic instability defined as cardiac index <2.0 l/min/m2 or systolic blood pressure <90mmHg or need for inotropic support or any mechanical circulatory support
* Left ventricular ejection fraction <25%
* Intracardiac mass or thrombus
* Co-morbid medical or oncologic condition for which local heart team believes that survival beyond 2 years is unlikely
* Active substance abuse
* Suspected inability to adhere to follow-up
* Treatment with another investigational drug or other intervention, assessment of which has not completed the primary endpoint or that clinically interferes with the present study endpoints.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2028-11-15 (Estimated); Study Completion 2030-11-15 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality, valve re-intervention, hospitalizations and urgent visits for heart failure, or onset of ≥ 2+ MR (by transthoracic echocardiogram (TTE)) composite score. | 3 years post intervention
  All-cause mortality, valve re-intervention, hospitalizations/urgent visits for heart failure (without a blanking period), or onset of > 32+ MR (by transthoracic echocardiogram (TTE)) from randomization to a minimum of 3 years post intervention.
  Composite score will be expressed as a Z-score - The Z-Score is a statistical measurement of a score's relationship to the mean in a group of scores. A Z-score of 0 is equal to the mean, with negative numbers indicating values lower than the mean and positive values higher than the mean.

SECONDARY OUTCOMES:
Adequacy of MR correction | one year post intervention
  Adequacy of MR correction at one year post intervention, defined as < 2+ MR as assessed by TTE
Kansas City Cardiomyopathy Questionnaire (KCCQ) | up to 10 years post intervention
  Disease-specific quality of life as measured by the KCCQ at 6-month time intervals up to 5 years. KCCQ has 23 items that map to 7 domains: symptom frequency; symptom burden; symptom stability; physical limitations; social limitations; quality of life; and self-efficacy. The symptom frequency and symptom burden domains are merged into a total symptom score, which can be combined with the physical limitation domain to create a clinical summary score. All scores are scaled 0 to 100, with higher scores indicating better health outcome.
Procedure failure | End of procedure
  Procedure failure defined as residual moderately severe or severe (3+ or 4+/4+) MR at the end of the procedure, or conversion of a TEER to an open surgical repair or replacement, or conversion of a surgical mitral valve repair to a mitral valve replacement procedure.
Procedure failure | 10 years post randomization
  Procedure failure defined as residual moderately severe or severe (3+ or 4+/4+) MR at the end of the procedure, or conversion of a TEER to an open surgical repair or replacement, or conversion of a surgical mitral valve repair to a mitral valve replacement procedure.
All-cause mortality | 5 years post randomization
  All-cause mortality through 5 years post randomization
All-cause mortality | 10 years post intervention
  All-cause mortality from randomization through 10 years post intervention
Cardiovascular and non-cardiovascular mortality | 5 years post intervention
  Cardiovascular and non-cardiovascular mortality from randomization through 5 years post intervention
Cardiovascular and non-cardiovascular mortality | 10 years post intervention
  Cardiovascular and non-cardiovascular mortality from randomization through 10 years post intervention
Valve re-interventions | 5 years post intervention
  Valve re-interventions through 5 years post intervention
Valve re-interventions | 10 years post intervention
  Valve re-interventions through 10 years post intervention
Serious or protocol-defined adverse events | 5 years post intervention
  Serious or protocol-defined adverse events, including stroke, acute kidney injury (AKI), and renal failure, through 5 years
MR grade | up to 6 years post intervention
  Mitral Regurgitation (MR) grade as mild, moderate, or severe. (grade I-IV, with higher grade indicating poorer health outcomes.)
Left Ventricular Ejection Fraction (LVEF) | up to 6 years post intervention
  Left ventricular ejection fraction (LVEF) is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction.
Left Ventricular End Diastolic Dimension (LVEDD) | up to 6 years post intervention
  Left ventricular end diastolic dimension (LVEDD) is the diameter across the left ventricle of the heart at the end of diastole, that is, when the heart muscle is maximally relaxed, and usually corresponds to its largest diameter.
Left Ventricular End Systolic Dimension (LVESD) | up to 6 years post intervention
  Left ventricular end systolic dimension (LVESD) is the diameter across the left ventricle of the heart at the end of systole, that is, when the heart muscle is maximally contracted, and usually corresponds to its smallest diameter.
Left Ventricular End Diastolic Volume (LVEDV) | up to 6 years post intervention
  Left Ventricular end diastolic volume (LVEDV) is the volume of blood in the left ventricle at the end of the diastole or ventricular filling.
Left Ventricular End Systolic Volume (LVESV) | up to 6 years post intervention
  Left Ventricular end systolic volume (LVESV) is the volume of blood in the left ventricle at the end of the systolic ejection phase immediately before the beginning of diastole or ventricular filling.
Mitral valve gradient | up to 6 years post intervention
  The valve gradient is the difference in pressure on each side of the valve. When a valve is narrowed (a condition called stenosis), the pressure on the front of the valve builds up as blood is forced through the narrow opening. This causes a larger pressure difference between the front and back of the valve. The valve gradient can be used to determine the severity of the valve disorder.
Forward stroke volume | up to 6 years post intervention
  The forward stroke volume is the volume entering the aorta.
6 Minute Walk Test (6MWT) | up to 5 years post intervention
  Functional status as measured by the 6MWT at yearly time intervals over 5 years. 6MT - The distance covered over a time of 6 minutes
EuroQol- 5 Dimension (EQ-5D) | through 10 years post intervention
  Generic QoL as measured by the EuroQol-5D (EQ-5D). The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ- 5D index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Length of stay (LOS) | through 10 years post intervention
  Length of stay as measured by number of days hospitalized.
ICU days of index hospitalization | through 10 years post intervention
  Number of ICU days of index hospitalization
Number and reasons for readmissions | through 10 years post intervention
  Number and reasons for readmissions, including for valve re-intervention and readmissions/urgent visits for heart failure
Cost | through 10 years post intervention
  Costs associated with the index hospitalization as well as follow-up readmissions will be measured.
Cost-effectiveness | through 10 years post intervention
  A cost-effectiveness analysis (CEA) comparing cumulative costs and quality-adjusted life years (QALYs) of transcatheter edge-to-edge repair vs surgical repair will be performed from U.S., Canadian, German and United Kingdom health care sector perspectives according to national guidelines.
Number of participants with stroke with disability | 30 days post-intervention
  Stroke with disability is defined as a modified Rankin score of ≥ 2 and/or major bleeding (BARC Type 3b, 3c and 5) by 30 days post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Chikwe, MD, Study Director — Cedars Sinai; Martin Leon, MD, Study Director — Columbia University; Patrick O'Gara, MD, Study Director — Brigham and Women's Hospital
Locations (61):
- United States (24):
  - Keck Hospital of the University of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Ochsner Clinic, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Saint Luke's Hospital of Kansas City/MidAmerica Heart and Lung Surgeons, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - Weill Cornell Medicine/ New York-Presbyterian Hospital, New York, New York
  - Northwell Health, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor, Scott and White, Dallas, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
- Canada (5):
  - University of British Columbia, Providence Health Care, St. Paul's Hospital, Vancouver, British Columbia
  - London Health Sciences, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Unity Health Toronto (St. Michael's Hospital), Toronto, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Laval University), Québec, Quebec
- Germany (15):
  - Universitätsklinikum Köln, Cologne, Berlin-kölnische Allee
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Kerckhoff Klinik Bad Nauheim, Bad Nauheim
  - Schüchtermann-Klinik Bad Rothenfelde, Bad Rothenfelde
  - Deutsches Herzzentrum der Charité, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Klinik St. Georg Hamburg, Hamburg
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Herzzentrum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - Deutsches Herzzentrum München, München
- Spain (4):
  - Hospital Alvaro Cunqueiro, Vigo, Galacia
  - Hospital Clinic De Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Central de Asturias, Oviedo
- United Kingdom (13):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge, England
  - The Leeds Teaching Hospitals NHS Trust, Leeds, England
  - St. Thomas Guy's and St Thomas' NHS Foundation Trust, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Royal Brompton and Harefield Guy's and St Thomas' NHS Foundation Trust, London, England
  - Manchester University NHS Foundation Trust, Manchester, England
  - University Hospitals Sussex NHS Foundation Trust, Worthing, West Sussex
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Golden Jubilee University National Hospital, Clydebank
  - Oxford University Hospitals NHS Foundation Trust, Headington
  - Barts Health NHS Trust, London
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - South Tees Hospital NHS Foundation Trust, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified study data sets must be submitted to the designated NHLBI Program Official no later than 3 years after the end of the clinical activity (final patient follow-up, etc.) or 2 years after the main paper of the trial has been published, whichever comes first. Data are prepared by the study coordinating center and sent to the designated PO for review prior to release.
Access Criteria: Anyone who wishes to access the data. Any purpose. Data are available indefinitely at link included in the URL field below.
URL: https://biolincc.nhlbi.nih.gov/studies/

REFERENCES:
- See also: PRIMARY Ancillary Substudy — https://clinicaltrials.gov/study/NCT07103733